CLINICAL TRIAL: NCT00046878
Title: Phase 2 Trial of BCNU Plus O6-Benzylguanine (NSC 637037) in the Treatment of Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Carmustine and O(6)-Benzylguanine in Treating Patients With Newly Diagnosed Supratentorial Glioblastoma Multiforme
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 3318; DUMC-3318-01-12; NCI-5632; CDR0000256332 (Other: NCI)
Record Dates: First submitted 2002-10-03; First posted 2003-08-11 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — O(6)-benzylguanine; Carmustine

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: carmustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. O(6)-benzylguanine may increase the effectiveness of carmustine by making tumor cells more sensitive to the drug.

PURPOSE: Phase II trial to study the effectiveness of combining carmustine with O(6)-benzylguanine in treating patients who have newly diagnosed supratentorial glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of carmustine and O6-benzylguanine in patients with newly diagnosed supratentorial glioblastoma multiforme not requiring immediate radiotherapy.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive O6-benzylguanine IV over 1 hour followed approximately 1 hour later by carmustine IV over 1 hour on day 1. Treatment repeats every 6 weeks for a maximum of 3 courses in the absence of disease progression or unacceptable toxicity. Patients are then referred for radiotherapy. Patients who demonstrate tumor response after completion of the third course of chemotherapy receive 6 additional courses after completion of radiotherapy.

PROJECTED ACCRUAL: A total of 19-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed supratentorial glioblastoma multiforme not requiring immediate radiotherapy
* Measurable residual disease on a contrast-enhanced MRI or CT scan (for patients with a medical contraindication for MRI) with a baseline scan obtained at the corticosteroid dose the patient is receiving on the day of treatment

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin greater than 10 g/dL

Hepatic

* Bilirubin normal
* SGOT no greater than 2.5 times upper limit of normal

Renal

* Creatinine no greater than 1.5 mg/dL
* BUN no greater than 25 mg/dL

Pulmonary

* DLCO greater than 75% predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics
* Concurrent corticosteroids allowed if on stable dose for 3 days before study

Radiotherapy

* See Disease Characteristics

Surgery

* No more than 28 days since prior surgical resection or biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute